CLINICAL TRIAL: NCT05183776
Title: Clinical Validation of a Fractional Administration Device for Holmium-166 Microspheres During Selective Internal Radiation Therapy in Patients With Liver Tumours
Brief Title: Clinical Validation of a Fractional Administration Device for Holmium-166 SIRT
Acronym: CONTROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONTROL
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Liver Cancer; Liver Metastasis Colon Cancer; Primary Liver Cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study patients (Experimental): study patients will receive holmium radioembolization using a novel administration device.
  Interventions: Device: Fractional administration device

INTERVENTIONS:
Device: Fractional administration device — The novel fractional administration device enable the administration of the microspheres in fractions determined by the user. For this study, 5 fractions of 20% will be administered and validated using MRI.

SUMMARY:
To investigate the in vivo performance and safety of a novel medical device for the injection of holmium-166 microspheres during radioembolization. The main potential advantage of this device is that it allows for injection of a during treatment determined dose, which is not possible with the current administration tool.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of hepatocellular carcinoma or liver metastases originating from colorectal cancer.
2. At least one lesion of ≥10 mm in the longest diameter on contrast-enhanced MRI or contrast-enhanced CT
3. Patient is eligible for SIRT as determined by the tumour board (in Dutch: MDO)
4. Patient has a life expectancy of 12 weeks or longer
5. Patient has a WHO performance score of 0-2

Exclusion Criteria:

1. Significant extrahepatic disease (2x sum of diameters of lesions outside the liver > sum of lesions inside the liver)
2. Radiation therapy, chemotherapy or major surgery within 4 weeks before treatment
3. Serum bilirubin > 2.0 x the upper limit of normal
4. ALAT, ASAT, alkaline phosphatase (AF) > 5x the upper limit of normal
5. Glomerular filtration rate (GFR-MDRD) <35 ml/min
6. Leukocytes <4.0 * 109/L or platelet count <60 * 109/L
7. Significant heart disease that in the opinion of the physician increases the risk of ventricular arrhythmia.
8. Pregnancy or breast feeding
9. Disease with increased chance of liver toxicity, such as primary biliary cirrhosis or xeroderma pigmentosum
10. Patients ineligible to undergo MR-imaging (claustrophobia, metal implants, etc)
11. Portal vein thrombosis of the main branch (more distal branches are allowed)
12. Evidence of clinically relevant, untreated grade 3 portal hypertension
13. Untreated, active hepatitis
14. Body weight > 150 kg (because of maximum table load)
15. Severe allergy for i.v. contrast (Iomeron, Dotarem and/or Primovist)
16. Lung shunt > 30 Gy, as calculated using scout dose holmium-166 SPECT/CT
17. Uncorrectable extrahepatic deposition of scout dose activity. Activity in the falciform ligament, portal lymph nodes or gallbladder are accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Validation of a fractional administration device for holmium radioembolization | 3 months after treatment
  The device will be valid if the administered fractions can be quantified on MRI with a maximal deviation of 15%.
Safety of a fractional administration device for holmium radioembolization | 6 months after treatment
  The safety of the device will be determined by monitoring the (S)AE's and (S)ADE's

SECONDARY OUTCOMES:
Accurate dosimetry based on MRI and SPECT imaging of holmium-166. | 6 months after treatment
  To perform dosimetry based on MRI and SPECT imaging of holmium-166 and correlate this to tumour response

CONTACTS AND LOCATIONS:
Overall Officials: Frank Nijsen, PhD., Principal Investigator — Associate professor
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Participant data will be available upon reasonable request